CLINICAL TRIAL: NCT03433677
Title: A Prospective, Randomized, Double-Blind, Crossover Comparison Evaluating Compatibility and Safety of LY900014 and Insulin Lispro With an External Continuous Subcutaneous Insulin Infusion System in Adult Patients With Type 1 Diabetes (PRONTO-Pump)
Brief Title: A Study of LY900014 and Insulin Lispro With an External Continuous Subcutaneous Insulin Infusion System in Adult Participants With Type 1 Diabetes
Acronym: PRONTO-Pump
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 16908; I8B-MC-ITSI (Other: Eli Lilly and Company); 2017-002374-39 (EudraCT Number)
Record Dates: First submitted 2018-02-09; First posted 2018-02-14 (Actual); Results first posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Diabetes Type 1
Keywords: insulin pump
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY900014 (Experimental): 100 units per milliliter (U/mL) LY900014 administered by individualized, continuous, subcutaneous insulin infusion (CSII)
  Interventions: Drug: LY900014
- Insulin Lispro (Experimental): 100 U/mL insulin lispro (Humalog®) administered by individualized CSII
  Interventions: Drug: Insulin lispro

INTERVENTIONS:
Drug: LY900014 — Administered by CSII
  Other Names: Ultra-Rapid Lispro
  Arms: LY900014
Drug: Insulin lispro — Administered by CSII
  Other Names: Humalog
  Arms: Insulin Lispro

SUMMARY:
The purpose of this study is to evaluate the compatibility and safety of LY900014 and insulin lispro with an external continuous subcutaneous insulin infusion system in adult participants with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 1 diabetes and have been using insulin continuously for at least 12 months.
* Using an insulin pump with 'rapid-acting insulin' for at least 6 months and using the same rapid-acting insulin for at least the past 30 days.
* Have experience using Continuous Glucose Monitoring (CGM) or Flash Glucose Monitoring (FGM) for at least 60 days during the past 12 months.
* Have hemoglobin A1c values ≤8.5%, as determined by the central laboratory at screening.
* Have a body mass index (BMI) of ≤35 kilograms per meter squared at screening.
* Have been using the MiniMed 530G or 630G (US) or the MiniMed 640G (EU) insulin pump for at least the past 30 days.

Exclusion Criteria:

* Have had more than 1 emergency treatment for very low blood glucose in the last 6 months.
* Have had more than 1 emergency treatment for poor glucose control (hyperglycemia or diabetic ketoacidosis) in the last 6 months.
* Have significant insulin resistance defined as having received a total daily dose of insulin >1.2 units per kilogram (U/kg) at screening, as determined by the average total daily insulin dose over the 3 days prior to screening divided by weight in kilograms based on investigator review of the participant's pump history.
* Have significant lipohypertrophy, lipoatrophy, or scars within the subcutaneous tissue in areas of infusion or have a history of abscess at an infusion site within the last 90 days prior to screening.
* Are receiving any oral or injectable medication intended for the treatment of diabetes mellitus other than rapid-acting analog insulin via CSII in the 90 days prior to screening. Occasional pen or syringe injection of insulin is allowed, for example, due to pump malfunction or unexplained hyperglycemia not responsive to pump correction bolus.
* Taking certain diabetes medications that are not allowed for study participation.
* Have major problems with heart, kidneys, liver, or have a blood disorder.
* Have had or are now being treated for certain types of cancer that prevents study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2018-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: 1-877-CTLILLY (1-877-285-4559) Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (3):
  - Valley Research, Fresno, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Atlanta Diabetes Associates, Atlanta, Georgia
- Spain (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Seville

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of LY900014 and Insulin Lispro With an External Continuous Subcutaneous Insulin Infusion System in Adult Participants With Type 1 Diabetes (PRONTO-Pump) — https://www.lillytrialguide.com/en-US/studies/type-1-diabetes/ITSI#?postal=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2-period crossover with no washout between periods and a 4 week safety follow-up.
Groups:
- Sequence 1 (LY900014/Insulin Lispro): 1. 100 U/mL LY900014 administered by continuous subcutaneous insulin infusion (CSII) for six weeks
  2. 100 U/mL insulin lispro (Humalog®) administered by CSII for six weeks with no washout between periods
- Sequence 2 (Insulin Lispro/LY900014): 1. 100 U/mL insulin lispro (Humalog®) administered by CSII for 6 weeks
  2. 100 U/mL LY900014 administered by continuous subcutaneous insulin infusion (CSII) for six weeks with no washout between periods
Period: Period 1
Arm/Group | Sequence 1 (LY900014/Insulin Lispro) | Sequence 2 (Insulin Lispro/LY900014)
Started | 24 | 25
Received at Least 1 Dose of Study Drug | 24 | 25
Completed | 23 | 25
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0
Period: Period 2
Arm/Group | Sequence 1 (LY900014/Insulin Lispro) | Sequence 2 (Insulin Lispro/LY900014)
Started | 23 | 25
Received at Least 1 Dose of Study Drug | 23 | 25
Completed | 22 | 24
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 (LY900014/Insulin Lispro) | Sequence 2 (Insulin Lispro/LY900014) | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.50 (12.47) | 36.72 (10.37) | 39.55 (11.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 12 | 11 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 23 | 25 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 23 | 25 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 11 | 21
  Spain | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Rate of Infusion Set Failures
Description: Infusion set failure events are defined as premature infusion set changes, due to a pump occlusion alarm OR due to unexplained hyperglycemia with blood glucose (SMBG) >250 milligrams per deciliter (mg/dL) (13.9 millimoles per liter [mmol/L]) that does not decrease within 1 hour following a correction bolus delivered via the pump during the 6 week treatment period. Aggregate rate was calculated for each participant as the total number of events while the participant is on study treatment divided by the days of exposure [last dose date and time -first dose date and time -duration of pump or treatment interruption] times 30.
Time Frame: 6 Weeks
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: events per 30 participant days
Groups:
- Insulin Lispro (Humalog®): 100 U/mL insulin lispro (Humalog®) administered by CSII
- LY900014: 100 U/mL LY900014 administered by continuous subcutaneous insulin infusion (CSII)
Arm/Group | Insulin Lispro (Humalog®) | LY900014
Number analyzed (Participants) | 48 | 49
events per 30 participant days | 0.05 | 0.03
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog®) vs LY900014; Test type: Superiority; p = 0.375, Wilcoxon signed-rank test; Median Difference (Final Values) = 0.00, 95% CI 2-sided [0.00 to 0.00]

2. Secondary Outcome: Percentage of Participants With at Least 1 Event of Infusion Set Failure
Description: Infusion set failures are defined as premature infusion set changes, due to a pump occlusion alarm OR due to unexplained hyperglycemia with blood glucose (SMBG) >250mg/dL (13.9 mmol/L) that does not decrease within 1 hour following a correction bolus delivered via the pump.
Time Frame: 6 Weeks
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Lispro (Humalog®) | LY900014
Number analyzed (Participants) | 48 | 49
percentage of participants | 6.3 | 4.1
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog®) vs LY900014; Test type: Superiority; p = 0.468, Prescott's Exact test

3. Secondary Outcome: Rate of Premature Infusion Set Changes
Description: Rate of premature infusion set changes.
Time Frame: 6 Weeks
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: events per 30 participant days
Arm/Group | Insulin Lispro (Humalog®) | LY900014
Number analyzed (Participants) | 48 | 49
events per 30 participant days | 0.78 | 1.13
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog®) vs LY900014; Test type: Superiority; p = 0.028, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Time Interval Until Infusion Set Change
Description: Time interval until infusion set change reflects the time interval in hours until infusion set change from first to last dose. MMRM model for post-baseline measures: Variable = Baseline + Period + Sequence + Strata(Region + Historical Use of SmartGuard/Threshold Suspend + HbA1c(<=7.3%, >7.3%)) + Treatment (Type III sum of squares).
Time Frame: 6 Weeks
Population: All randomized participants who received at least 1 dose of study drug and non-missing baseline value and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Insulin Lispro (Humalog®) | LY900014
Number analyzed (Participants) | 46 | 47
hours | 76.1 (1.52) | 74.3 (1.51)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog®) vs LY900014; Test type: Superiority; p = 0.304, Mixed Models Analysis; LSMean Difference = -1.8, 95% CI 2-sided [-5.3 to 1.7]

5. Secondary Outcome: Ratio of Bolus/Total Insulin Dose
Description: The bolus and total insulin doses for each visit was calculated as the mean of the doses for the last 3 days prior to the visit date that are entered in the eCRF. The bolus/total ratio was derived as the bolus dose divided by the total insulin dose at each visit.
Time Frame: 6 Weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: percentage of total insulin dose
Arm/Group | Insulin Lispro (Humalog®) | LY900014
Number analyzed (Participants) | 47 | 46
percentage of total insulin dose | 46.6 (1.17) | 44.2 (1.17)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog®) vs LY900014; Test type: Superiority; p = 0.057, Mixed Models Analysis; LSMean Difference = -2.4, 95% CI 2-sided [-4.8 to 0.1]

6. Secondary Outcome: Interstitial Glucose Reduction Rate From Hyperglycemia Following a Non-Meal-Related Correction Bolus Delivered Via the Pump
Description: Interstitial glucose reduction rate (glucose reduction [mg/dL] per minute) within 4 hours following a non-meal-related correction bolus via the pump, from hyperglycemia (interstitial glucose >180 mg/dL [10 mmol/L]) to recovery (interstitial glucose ≤180 mg/dL).
Time Frame: 6 Weeks
Population: All randomized participants who received at least 1 dose of study drug and non-missing baseline value and at least one non-missing post-baseline value of the response.
Measure: Least Squares Mean (Standard Error); unit: mg/dL/min
Arm/Group | Insulin Lispro (Humalog®) | LY900014
Number analyzed (Participants) | 37 | 37
mg/dL/min | 0.71 (0.062) | 0.82 (0.063)
Statistical Analysis 1: Comparison: Insulin Lispro (Humalog®) vs LY900014; Test type: Superiority; p = 0.177, Mixed Models Analysis; LSMeans = 0.11, 95% CI 2-sided [-0.05 to 0.27] — LSMean Difference

7. Secondary Outcome: Number of Participants With Severe Hypoglycemic Events
Description: Number of participants with severe hypoglycemic events. Severe hypoglycemia was defined as participants with an altered mental status and could not assist in their own care, may have been semiconscious or unconscious, or experienced coma with or without seizures, and the event required assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. Blood glucose measurements may not have been available during such an event, but neurological recovery attributable to the restoration of BG concentration to normal was considered sufficient evidence that the event was induced by a low BG concentration (BG ≤70 mg/dL [3.9 mmol/L]).
Time Frame: 6 Weeks
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Insulin Lispro (Humalog®) | LY900014
Number analyzed (Participants) | 48 | 49
participants | 1 | 1

ADVERSE EVENTS:
Time Frame: up to 12 weeks
Description: All randomized participants who received at least 1 dose of study drug.
Groups:
- LY900014: LY900014 administered by continuous subcutaneous insulin infusion (CSII)
- Insulin Lispro (Humalog®): Insulin lispro (Humalog®) administered by CSII
Arm/Group | LY900014 | Insulin Lispro (Humalog®)
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/48
Serious Adverse Events (participants affected / at risk) | 1/49 | 1/48
Other Adverse Events (participants affected / at risk) | 18/49 | 6/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY900014 (N=49) | Insulin Lispro (Humalog®) (N=48)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY900014 (N=49) | Insulin Lispro (Humalog®) (N=48)
Infusion site pain (General disorders) | 9 (11) | 2 (2)
Infusion site reaction (General disorders) | 9 (36) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-01-12): https://cdn.clinicaltrials.gov/large-docs/77/NCT03433677/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT03433677/SAP_001.pdf